CLINICAL TRIAL: NCT02900469
Title: Pre-surgical Evaluation of Denosumab in Patients With Operable Invasive Breast Cancer
Brief Title: Presurgical Trial of Denosumab in Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s14-01311
Record Dates: First submitted 2016-08-29; First posted 2016-09-14 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
Keywords: RANK; RANKL
MeSH Terms: conditions — Breast Neoplasms | interventions — Denosumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Denosumab & surgery (Experimental): denosumab: 120 mg subcutaneous injection
  Surgery: 2-4 weeks after denosumab
  Interventions: Biological: denosumab; Procedure: Surgery

INTERVENTIONS:
Biological: denosumab — denosumab: 120 mg subcutaneous injection
  Other Names: Xgeva
Procedure: Surgery — Surgery: approximately 2-4 weeks after dosing of denosumab

SUMMARY:
The purpose of this study is to determine whether one dose of denosumab can lead to changes in the tumor, which may decrease the ability of tumor to spread.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among women, affecting one in eight women, and is the second leading cause of mortality from cancer. Bone metastases are a frequent complication of breast cancer, and the mechanism of breast cancer metastases to bone is an ongoing area of research.. Receptor activator of NF-kB (RANK) and its ligand (RANKL) have been identified and characterized for its role in bone remodeling. RANKL is a member of the tumor necrosis factor (TNF) family of cytokines that binds to its receptor RANK to control osteoclast differentiation, activation, and survival. RANK protein expression is not only found on osteoclasts and dendritic cells but also on T cells and mammary epithelial cells. RANK and RANKL is important for lymph node and thymus formation as well as lactating mammary gland development during pregnancy. Furthermore, the RANK/RANKL axis has been linked to progestin driven breast carcinomas and bone metastases.

RANK is expressed in 6-57% of invasive human breast cancers (depending upon the parameters for defining positivity and antibodies utilized for immunohistochemistry (IHC)), and RANKL driven hormone (progesterone -dependent proliferation, survival, and nonproliferative expansion of mammary stem cells may contribute to breast cancer initiation, progression, and recurrence.

We hypothesize that denosumab can inhibit RANKL signaling in early breast tumors which express RANK, inhibiting pro-metastatic mechanisms and reducing immunosuppression in the tumor microenvironment. This will be tested in a pre-surgical clinical trial (Phase 0) to evaluate and select the pharmacodynamics markers of RANKL inhibition in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed invasive breast cancer (stages I-III) who have undergone core needle biopsy (clinically or radiographically at least T1c to allow adequate residual cancer tissue at surgery) and will be scheduled for surgical resection (i.e. segmental excision or mastectomy).
* Archival tissue freshly cut from core biopsy must be available; patients who had a diagnostic core biopsy at an outside institution are eligible as long as it is confirmed that tumor specimens in paraffin blocks (preferred) or ≥ 25 unstained slides, with an associated pathology report, are available.
* Female, Age ≥18 years (pre or postmenopausal).
* Signed informed consent
* Serum calcium or albumin-adjusted serum calcium ≥2.0mmol/L (8.0mg/dL) and ≤ 2.9 mmol/L (11.5mg/dL)
* Patients with reproductive potential must be willing to use, in combination with her partner, 2 acceptable methods of effective contraception or practice sexual abstinence throughout the study and continue for 5 months after study duration. Subjects who are surgically sterile (eg, history of bilateral tubal ligation, hysterectomy) or whose sexual partner is sterile (eg, history of vasectomy) are not required to use additional contraceptive measures.

Exclusion Criteria:

* Consideration for neoadjuvant therapy
* Serious infections including a history of active Hepatitis B, Hepatitis C or HIV
* Subject has known sensitivity to any of the products to be administered during the study (e.g.., mammalian derived products, calcium, or vitamin D)
* Subject is pregnant or breast feeding, or planning to become pregnant/breastfeed while on study through 5 months after the end of treatment
* Patients have prior history or current evidence of osteonecrosis or osteomyelitis of the jaw, evidence of untreated local gum or oral infection, or non-healed dental or oral surgery
* Patients with active dental or jaw conditions which require oral surgery/dental procedures, including tooth extraction for the course of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-10; Primary Completion 2019-12-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic markers of RANKL inhibition determination | Change from baseline RANKL inhibition determination at one month
  Immunohistochemical analyses (IHC) of RANK and RANKL protein expression will be performed by Clarient Diagnostics Services Inc., Aliso Viejo, CA using prototype assays developed and optimized by Dako on their automated staining platform

SECONDARY OUTCOMES:
Frequency of RANK and RANKL protein expression (by IHC) in operable breast cancer using Immunohistochemical analyses (IHC) | Change from baseline frequency of RANK and RANKL protein expression at one month
  Immunohistochemical analyses (IHC) of RANK and RANKL protein expression will be performed by Clarient Diagnostics Services Inc., Aliso Viejo, CA using prototype assays developed and optimized by Dako on their automated staining platform

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Adams, MD, Principal Investigator — NYU Perlmutter Cancer Center
Locations (1):
- NYU Perlmutter Cancer Center, New York, New York, United States